CLINICAL TRIAL: NCT06713603
Title: Technology Assisted Motivational Interviewing Randomized Controlled Trial
Brief Title: Technology Assisted Motivational Interviewing
Acronym: TAMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-41634; T34IR7967 (Other Grant/Funding Number: TRDRP)
Record Dates: First submitted 2024-10-30; First posted 2024-12-03 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Smoking; Smoking Cessation
Keywords: smoking; quit smoking; motivational interviewing; chatbot; cessation; coach; motivation; quit plan
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into intervention or usual care.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology Assisted Motivational Interviewing (TAMI) (Experimental): Individuals randomized to TAMI will interact with the fully automated, web-based MI-chatbot for the 6-month study period. Patients who continue to smoke will receive up to two text messages per week with the chatbot URL link to initiate additional conversations always beginning with an assessment of readiness to change but "remembering" prior conversations much like a clinician. Individuals in the preparation stage will move directly to EBP education, tailoring a quit plan and boosting both self-efficacy and outcome expectancies. Patients with sufficient confidence will be encouraged to set a quit date. Patients will be encouraged to include their PCP and/or state quitline. TAMI will provide support proximal to the quit date including guidance through common obstacles. TAMI will check back to assess treatment initiation, treatment sustainment (and/or cessation), or relapse. Patients who are unable to quit (or who relapse) will be encouraged to restart conversations with TAMI.
  Interventions: Behavioral: TAMI Coach
- Usual Care (No Intervention): Individuals randomized to the Usual Care (UC) condition will receive a detailed educational handout on the health risks associated with smoking and information on Evidence Based Practice's (EBP) for cessation using the standard "Kick-It California" materials. Additional materials and referral resources regarding depression, stress, and other common barriers will be provided to all UC participants. Any UC individual can choose to quit at any time but they will not have access to TAMI. While this is not an "active" treatment condition, the handout and recurring assessments (at 3 and 6mo) may serve as reminders about the importance of quitting and may assist with finding support for co-occurring conditions or social needs.

INTERVENTIONS:
Behavioral: TAMI Coach — The investigators address the problems of intrinsic motivation, Evidence Based Practice (EBP) education, and referral tailoring using a digital-coaching intervention that 1) promotes readiness to change, 2) educates and builds confidence about EBP's, and 3) creates a tailored quit plan sensitive to social obstacles and needs.
  Arms: Technology Assisted Motivational Interviewing (TAMI)

SUMMARY:
Building on our successful pilot work to develop a Motivational Interviewing (MI)-capable chatbot and cessation coach, the investigators propose to address the problems of intrinsic motivation and social barriers to smoking cessation by evaluating a highly scalable and easily accessible digital-coaching intervention that 1) promotes readiness to change using a technology-assisted MI (TAMI) chatbot, 2) provides compelling and accessible multilingual education about smoking cessation tools, and 3) develops a tailored quit plan addressing social barriers to treatment initiation and sustainment.

ELIGIBILITY:
Inclusion Criteria:

* A current Primary Care Provider patient
* Age 18 or older
* Smoke at least 1 cigarette per day for the past 7 consecutive days (and at least 100 lifetime)
* Have a digital device (phone, laptop, tablet)
* Moderately proficient in English
* Able to participate for 6-month trial

Exclusion Criteria:

* Current participation in a smoking cessation program
* Current use of Nicotine Replacement Therapy or smoking cessation pharmacotherapy
* Cognitive impairment that would preclude informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical verification of smoking abstinence | 6-month
  The primary clinical outcome is 7-day point prevalence abstinence (PPA) from smoking at 6-months. Abstinence will be biochemically verified with salivary cotinine.
  To maximize the validity of our primary abstinence outcome, the investigators will require any participant in who reports abstinence at 6-month to complete salivary cotinine bio-verification using a mailed, commercially available test kit. Participants will be instructed to electronically send two photos - one of them giving a saliva sample and the other with the test results. Recent reviews of biochemical verification strategies have validated this methodology. People with at least 10 ng/ml cotinine in their saliva will be considered smokers. The investigators will ask participants to report any Nicotine Replacement Therapy use or vaping to identify false positives.

SECONDARY OUTCOMES:
Self reported smoking abstinence | 3-month
  Self-reported point prevalence abstinence (PPA) from smoking at 3-month
Smoking reduction | Baseline, 3-month, 6-month
  Self reported smoking reduction (# cigs, >50% reductions, and # quit attempts). Change = (score at time point - score at baseline)
Readiness to quit | Baseline, 3-month, 6-month
  Self reported changes in readiness to quit, and treatment initiation and sustainment. Possible scores range from 1 (not at all) to 10 (totally ready). Change = (score at time point - score at baseline)
Smoking cessation outcome expectations | Baseline, 3-month, 6-month
  Self reported smoking cessation outcome expectations measuring how serious would the health consequences be if the participant developed a smoking-related disease. Possible scores range from 1 (Not at all) to 5 (Extremely serious). Change = (score at time point - score at baseline)
Self-efficacy | Baseline, 3-month, 6-month
  The Smoking Self-Efficacy Questionnaire (SEQ-12) is a validated, self reported 12-item instrument that measures the confidence of current and former smokers in their ability to abstain from smoking in certain social or emotional situations. The SEQ-12 has two subscales measuring confidence in ability to refrain from smoking when facing internal stimuli (e.g., feeling depressed) and external stimuli (e.g., being with smokers). Possible scores range from 1 (not at all sure) to 5 (absolutely sure). The scores for each question are added together. A higher score indicates greater self-efficacy. Change = (score at time point - score at baseline)
Chatbot engagement and usage | Baseline, 3-month, 6-month
  The Mobile App Rating Scale is a validated, self reported instrument measuring app quality across four dimensions: engagement, functionality, aesthetics and information quality. Possible scores range from 1 (not at all useful) to 4 (very useful. Change = (score at time point - score at baseline)
Digital Health Literacy survey | Baseline, 3-month, 6-month
  The Digital Health Literacy instrument is a validated, self-reported 8-item instrument measuring digital health literacy in general adult populations. Possible scores range from 1 (strongly disagree) to 5 (strongly agree). Change = (score at time point - score at baseline)
AHC Screening Tool | Baseline, 3-month, 6-month
  The Accountable Health Communities screening tool is a validated, self reported 10-item instrument assessing social needs. Change = (score at time point - score at baseline)
Bayliss Disease Burden | Baseline, 3-month, 6-month
  Bayliss Disease Burden
  The Bayliss Disease Burden Morbidity Assessment is a validated, self-reported instrument serving as a subjective measure of comorbidity that incorporates an assessment of disease severity. Possible scores range from 1 (not at all) to 5 (a lot). Disease burden is defined as the number of self-identified comorbid conditions weighted by the degree to which each interfered with their daily activities. Change = (score at time point - score at baseline)
PHQ-8 | Baseline, 3-month, 6-month
  The Personal Health Questionnaire Depression Scale is a validated, self-reported 8-item instrument assessing symptoms of depression. Possible scores range from 0 (not at all) to 3 (nearly every day). The scores for each question are added together. A higher score indicates greater depression. Change = (score at time point - score at baseline)
Perceived Stress Scale | Baseline, 3-month, 6-month
  The Perceived Stress Scale is a validated, self-reported 10-item instrument assessing how stressful a person finds their life to be. Possible scores range from 0 (never) to 4 (very often). The scores for each question are added together. A higher score indicates greater perceived stress. Change = (score at time point - score at baseline)

OTHER OUTCOMES:
Demographics | Baseline, 6-month
  Self reported demographics
User experience and satisfaction | Baseline, 6-month
  The Working Alliance Inventory is a validated, self-reported 12 item instrument measuring three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. Possible scores range from 1 (seldom) to 5 (always).
  Change = (score at time point - score at baseline)
Treatment barriers/facilitators | 6-month
  Open feedback on treatment barriers/facilitators via 1:1 Exit Interviews

CONTACTS AND LOCATIONS:
Overall Officials: Jason Satterfield, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco General Hospital, San Francisco, California
  - UCSF Adult Primary Care Mt. Zion Clinic, San Francisco, California

IPD SHARING:
Plan to Share IPD: No
This project is funded by the UC Tobacco-Related Disease Research Program (TRDRP) and will use the data sharing platform required for that consortia.

REFERENCES:
- [Derived] Borsari B, Meacham MC, Saiyed A, Kanzaveli T, Tsvetovat M, Cheng J, Hargrave-Bouagnon AS, Mirzadegan IA, Omeragic F, Layton J, Satterfield J. Protocol for a randomized clinical trial to evaluate the effectiveness of a technology-assisted motivational interviewing (TAMI) chatbot on smoking cessation. Contemp Clin Trials. 2025 Dec;159:108111. doi: 10.1016/j.cct.2025.108111. Epub 2025 Oct 22. PMID 41135811